CLINICAL TRIAL: NCT02344121
Title: Intra- and Inter-fraction Changes in Radiation Therapy
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Eric Paulson, Associate Professor, Medical College of Wisconsin
Other Study IDs: 22316
Record Dates: First submitted 2014-12-05; First posted 2015-01-22 (Estimated); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation therapy plans for cancer patients who have completed treatment.

SUMMARY:
Analysis to quantify intra-fraction, inter-fraction and post-treatment changes in tumor target volumes and surrounding normal organs in radiation therapy.

DETAILED DESCRIPTION:
The accurate and detailed knowledge of the changes (e.g., anatomically/biologically intra- and inter-fraction changes) to be obtained from this study would allow the research team to determine how Adaptive Radiation Therapy (ART) should be performed for a given tumor site/type. Radiation oncologists then can choose a proper ART strategy for a given tumor type to account for the anatomic/biological intra- and inter-fraction changes, improving accuracy of radiation therapy delivery, and in turn reducing treatment related toxicities and/or improving tumor local control.

ELIGIBILITY:
Inclusion Criteria:

°Completed radiation therapy

Exclusion Criteria:

°Subjects who refuse voluntary participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients who have completed treatment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-01; Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-20 (Estimated)

PRIMARY OUTCOMES:
Changes of volumes from baseline of organs at risk during and after radiation therapy. | 2 years
  Changes of organs at risk volumes (cm^3) during and after radiation therapy.

SECONDARY OUTCOMES:
Changes of volumes from baseline or tumors during and after radiation therapy. | 2 years
  Changes of tumor volumes (cm^3) during and after radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Paulson, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No